CLINICAL TRIAL: NCT05690880
Title: ForeseeHome NRich Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Notal Vision Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FSH-R-C2022.001
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Foresee Home — The ForeseeHome Monitoring System, a non-significant risk device, is prescribed by eye care providers to patients as part of their clinical care. Notal Vision Monitoring Center (NVMC) is an independent diagnostic testing facility responsible for clinical monitoring of FSH data. The NVMC communicates with the patients (for training on the use of the device, troubleshooting of device issues, adherence monitoring, etc.) and with the patients' eyecare providers (for reporting FSH alerts, monitoring of clinical outcomes to assess device functionality and ongoing need for the device, etc.).

SUMMARY:
This registry will compare functional and structural data of progression of Intermediate AMD (iAMD) and conversion to neovascular AMD (NV-AMD) while monitored at home with the ForeseeHome Monitoring System (FSH) and during routine care with Spectral Domain Optical Coherence Tomography (SD-OCT) and to validate the predictive value of a non-NV-AMD FSH alerts.

DETAILED DESCRIPTION:
The participants include those actively monitoring on the FSH program which requires diagnosis of intermediate AMD and visual acuity of 20/60 or better that establish a valid baseline in at least one eye. The process of establishing a baseline is completed several weeks after setup of the device at home and initiation of testing. The aim of the registry is to collect data up to 20,000 patients on the ForeseeHome program for at least one year. The data will be collected for approximately a period of 5 years.

The registry will include clinics that provide direct care to the patients on the ForeseeHome device, and Notal Vision Monitoring Center. The registry aims to collect data from about 200 referring physicians.

The registry will include structural and functional data for the patients active on the ForeseeHome device. The details of data points to be collected are mentioned below.

Data from participating sites will be collected in a de-identified manner and collected in the registry. Patients will be assigned a patient ID and will be collected in a sequential manner from each site. No data shall be acquired outside standard of care. Not all data points for each patient are expected to be present. The following data points shall be shared in the registry:

From Notal Vision Monitoring Center

1. Patient ID, Date of Birth (DOB), gender, and testing eye From prescribing physician
2. Visual Acuity: Visual acuity as measured during regular examination, in a period when the patient is active on the ForeseeHome program, shall be shared in the registry. Maximum 2 visual acuity measurements shall be shared during one calendar year.
3. Structural OCT Images: OCT images (volume scans) acquired following a ForeseeHome alert shall be shared in the registry.
4. OCT Angiography (OCT-A) Images: OCT-A images acquired following a ForeseeHome alert shall be shared in the registry
5. Fluorescein Angiography (FA): FA images acquired following a ForeseeHome Alert visit shall be shared in the registry
6. Diagnosis of wet-AMD in case of ForeseeHome alert: The diagnosis related to status of patient's macular degeneration in both eyes shall be shared in the registry in case of an alert.
7. Status of the eye after exiting the ForeseeHome program regarding conversion to wet-AMD and its timing

ELIGIBILITY:
Inclusion Criteria:

* The participants include those actively monitoring on the FSH program which requires diagnosis of intermediate AMD and visual acuity of 20/60 or better that establish a valid baseline in at least one eye.

Exclusion Criteria:

* Patients that are unable to establish a baseline

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participants include those actively monitoring on the FSH program which requires diagnosis of intermediate AMD and visual acuity of 20/60 or better that establish a valid baseline in at least one eye. The process of establishing a baseline is completed several weeks after setup of the device at home and initiation of testing. The aim of the registry is to collect data up to 20,000 patients on the ForeseeHome program for at least one year. The data will be collected for approximately a period of 5 years.The registry will include clinics that provide direct care to the patients on the ForeseeHome device, and Notal Vision Monitoring Center. The registry aims to collect data from about 200 referring physicians.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
This registry will compare functional and structural data of progression of Intermediate AMD (iAMD) and conversion to neovascular AMD (NV-AMD) | 5 years
  This registry will compare functional and structural data of progression of Intermediate AMD (iAMD) and conversion to neovascular AMD (NV-AMD) while monitored at home with the ForeseeHome Monitoring System (FSH) and during routine care with SD-OCT and to validate the predictive value of a non-NV-AMD FSH alerts.

CONTACTS AND LOCATIONS:
Locations (1):
- NJ Retina, Toms River, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No